CLINICAL TRIAL: NCT03222349
Title: A Multicenter,Open Label Crossover Study to Assess the Pharmacokinetics and Safety of Diazepam Buccal Soluble Film (DBSF) in Pediatric Subjects With Epilepsy
Brief Title: Pharmacokinetics and Safety Study of Diazepam Buccal Film (DBF) in Pediatric Subjects With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aquestive Therapeutics (Industry)
Collaborators: Syneos Health (Other); Covance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 160325
Record Dates: First submitted 2017-07-12; First posted 2017-07-19 (Actual); Results first posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Epilepsy
Keywords: interictal state; ictal/peri-ictal state
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: This was a multicenter study comprised of 2 treatment periods with a minimum 14 days between the 2 treatment periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Interictal Period (Experimental): Each subject received a single dose of DBF based on the subject's age and weight.
  Interventions: Drug: Diazepam Buccal Film
- Ictal/Peri-ictal Period (Experimental): Each subject received a single dose of DBF based on the subject's age and weight.
  Interventions: Drug: Diazepam Buccal Film

INTERVENTIONS:
Drug: Diazepam Buccal Film — Subjects received a single DBF dose determined by age and body weight during the interictal state and during the ictal/peri-ictal period with at least 14 days washout between doses.
  Other Names: DBSF

SUMMARY:
Open-label study to assess the pharmacokinetics of a single diazepam buccal film (DBF) dose in 3 age cohorts of pediatric patients with epilepsy (age 2-5 years, age 6-11 years, and age 12-16 years). Subjects in the 6-11 years and 12-16 years age cohorts received a single DBF dose during the interictal period (Period A) and ictal/peri-ictal period (Period B) with at least 14 days washout between doses. Subjects in the age 2-5 years age cohort received a single DBF dose only during the ictal/peri-ictal period (Period B).

DETAILED DESCRIPTION:
This was a Phase 2 multicenter, open-label, two-way study conducted in male and female pediatric subjects (aged 2 to 16 years) with a clinical diagnosis of epilepsy who were scheduled to be admitted to an Epilepsy Monitoring Unit (EMU), a general clinical research center (GCRC), or similar facility for evaluation of seizures and who complied with all remaining protocol eligibility criteria. To ensure that 16 to 18 subjects would complete the study across 3 age ranges (2 to 5 years, 6 to 11 years, and 12 to 16 years), a minimum of 24 subjects were to be enrolled (8 in each age cohort).

Subjects in the 6 to 11 years and 12 to 16 years age cohorts received a single dose of DBF during the interictal period (Period A) and ictal/peri-ictal period (Period B) with at least 14 days washout between doses. Subjects in the age 2 to 5 years age cohort received a single dose of DBF only during the ictal/peri-ictal period (Period B). DBF was provided in a range of doses from 5 to 17.5 mg. The appropriate dose of DBF was assigned on the basis of age and weight using an interactive web response system during check-in.

Period A (interictal administration): Subjects were considered to be in an interictal state if an interval of at least 3 hours had elapsed since any clinically observable postictal signs or symptoms (from the last observed seizure) and the subject had been seizure-free over this period. Subjects on electroencephalogram (EEG) monitoring were to be considered to be in an interictal state if an interval of at least 3 hours had elapsed since there were any postictal electrical findings on EEG.

Period B (ictal/peri-ictal administration): For the purpose of this study, the ictal state was defined as an ongoing clinically observable seizure or seizure activity as verified via EEG. The peri-ictal state was defined clinically as the subject's immediate postictal state following a generalized tonic-clonic (GTC) seizure or focal seizure with impaired awareness, and within 5 minutes following the last clonic jerk. For subjects on EEG monitoring, the peri-ictal state was to be defined as less than 5 minutes after cessation of seizure activity as verified via EEG.

.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects meeting all of the following criteria may be included in the study:

1. Subjects have a clinical diagnosis of epilepsy (GTC seizures or focal seizures with impaired awareness) and were scheduled for admission to an Epilepsy Monitoring Unit (EMU), General Clinical Research Center (GCRC), or similar facility for evaluation.
2. Male and female subjects between 2 and 16 years of age, inclusive.
3. Subjects had a body weight of at least 6 kg and less than or equal to 111 kg.
4. Subjects had an average frequency of at least 1 clinically apparent seizure every 3 days or ≥10 clinically apparent seizures per month, with alteration of consciousness as documented by reliable subject report, personal seizure diary records, and/or by seizure diaries dispensed at screening and verified prior to study entry.
5. Female subjects of childbearing potential (i.e., were having periods, were not surgically sterile) must have had a negative serum pregnancy test (using Beta-hCG) at Screening and a negative urine pregnancy test on Study Day I prior to drug dosing. Female subjects of childbearing potential must have agreed to abstinence, have had a partner who was sterile, or have been practicing double barrier contraception or have been using an FDA-approved contraceptive (e.g., licensed hormonal or barrier methods) for greater than 2 months prior to screening visit, and must have committed to an acceptable form of birth control for the duration of the study and for 30 days after participation in the study.
6. Male subjects with a female sexual partner of childbearing potential must have agreed to abstinence or to practice adequate birth control during the study, including at least 1 barrier method such a condom, diaphragm, or spermicide for more than 2 months prior to the screening visit, and must have committed to an acceptable form of birth control for the duration of the study and for 30 days after participation in the study. Also, male subjects must have agreed not to donate sperm during the study and for 90 days after the follow-up visit.
7. Subjects were currently receiving at least one antiepileptic medication.
8. Subject's parent or legally authorized representative must have been willing and able to complete informed consent and HIPAA authorization. Subjects must have been willing to give assent as required by the Institutional Review Board (IRB).
9. Subject must have agreed to be available or subject's parent(s) or legally authorized representative(s) must have agreed to have the subject be available for both Treatment Periods and the Follow-up Visit, and must have been willing to comply with all required study procedures and adhere to all protocol requirements.
10. Subject or subject's parent(s) or legally authorized representative(s) must have been able to comprehend and be informed of the nature of the study, as assessed by the Investigator.

Exclusion Criteria:

Potential subjects meeting any of the following criteria were excluded from participating in the study:

1. Subjects with a progressive neurological disorder such as a brain tumor, demyelinating disease, or degenerative central nervous system (CNS) disease that was likely to progress in the 12 months after screening.
2. Subjects with respiratory failure (or is at risk for respiratory failure) or other severe cardiorespiratory disease with New York Heart Association Class Ill or IV functional status, or who required supplemental oxygen.
3. Female subjects who were lactating, had a positive serum pregnancy test (β-hCG) at screening, or had a positive urine pregnancy test at Check-in for treatment periods.
4. Subjects with psychiatric disease that in the Investigator's judgment would prevent the subject's successful completion of the study.
5. Subjects with recent history of suicide attempt (defined as an active, interrupted, or aborted attempt within the previous 5 years) or reported suicidal ideation in the previous 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale performed at the screening visit.
6. Subjects with known history or presence of any clinically significant hepatic (e.g., hepatic impairment), renal/genitourinary (renal impairment, kidney stones), psychiatric, dermatological, or hematological disease or condition, unless determined as not clinically significant by the Investigator or designee and confirmed by Sponsor via written communication prior to subject enrollment. Abnormal laboratory results considered clinically significant by the Investigator or designee were to be evaluated by the Investigator in consultation with the Medical Monitor.
7. Subjects with any clinically significant illness other than epilepsy within 30 days prior to study drug administration, as determined by the Investigator.
8. Subjects with any significant physical or organ abnormality or other condition that would interfere with study participation or constitute a safety risk in the judgment of the Investigator.
9. Subjects with any significant lesion of the oral cavity or having oral prophylactic or dental procedures within 30 days prior to study drug administration.
10. Subjects with a QT interval corrected by Fridericia's formula (QTcF) >450 ms for males or QTcF >470 ms for females on screening ECG unless determined as not clinically significant by the Investigator.
11. Subjects with a positive test result for any of the following drugs of abuse:

    amphetamines, cocaine, opiates, phencyclidine, or a positive breath alcohol test. Subjects who tested positive for tetrahydrocannabinol (THC) at screening were excluded unless the Investigator was able to affirm in writing that the use of a medical marijuana product was part of the subject's treatment plan as recommended by a physician for treatment of a medical condition. In such case, the subject was to be allowed to continue with screening, and the medical marijuana product was to be recorded as a concomitant medication.
12. Subjects with a known history or presence of any of the following:

    1. Substance abuse or dependence (including alcohol) within 1 year prior to first study drug administration
    2. Hypersensitivity or idiosyncratic reaction to diazepam, its excipients, sodium phosphates, and/or related substances, e.g., benzodiazepines
    3. Glaucoma (open or acute narrow angle)
    4. Severe allergic reactions (e.g., anaphylactic reactions, angioedema) to investigational product and excipients
13. Subjects who had participated in another clinical trial or who had received an investigational drug within 30 days prior to study drug administration or 5 half-lives of the investigational drug-whichever was the longer period.
14. Subjects with presence of mouth jewelry, dentures, oral implants, braces, or piercings in the mouth or tongue that, in the opinion of the Investigator, would have been likely to interfere with successful completion of the dosing procedure.
15. Subjects with a blood or plasma donation within 30 days prior to screening.
16. Subjects not willing or unable to tolerate blood draws.
17. Consumption of alcohol within 48 hours before dosing; or food or beverages containing grapefruit, star fruit, Seville oranges, and/or pomelo, or their derived products (e.g., fruit juice) within 10 days prior to study drug administration.
18. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome (CYP) 450 enzymes (e.g., cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem, or HIV antivirals) and strong inducers of CYP enzymes (e.g., glucocorticoids, St. John's Wort, or rifampicin), in the previous 30 days prior to study drug administration. (Barbiturates, carbamazepine, phenytoin, and other enzyme-modifying antiepileptic drugs (AEDs) that were medically needed were permitted.)
19. Use of any monoamine oxidase (MAO) inhibitors (e.g., phenelzine, tranylcypromine ), and/or phenothiazines (chlorpromazine) within 30 days prior to first study drug administration.
20. Employee or immediate relative of an employee of Aquestive Therapeutics, any of its affiliates or partners, or Syneos Health.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Slatko, Study Director — Aquestive Therapeutics
Locations (10):
- United States (10):
  - University of Arizona, Tucson, Arizona
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Children's St. Peters University Hospital, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester, Rochester, New York
  - Onsite Clinical Solutions LLC, Charlotte, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Dell Children's Medical Center, Austin, Texas
  - Austin Epilepsy Care Center, Austin, Texas
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned enrollment was 24 male and female subjects with 8 subjects in each of 3 age ranges (2 to 5 years, 6 to 11 years, and 12 to 16 years) with a clinical diagnosis of epilepsy (generalized tonic clonic seizures or focal seizures with impaired awareness) currently receiving at least one epileptic medication who were scheduled for admission to an Epilepsy Monitoring Unit (EMU), General Clinical Research Center (GCRC), or similar facility for evaluation.
Pre-assignment Details: A total of 24 subjects were enrolled and received at least 1 dose of study drug based on age and weight during the interictal and the ictal/peri-ictal period in either order as determined by seizure occurrence.
Groups:
- Interictal State, Then Ictal/Peri-ictal State: The interictal state was defined as a period of time during which 3 hours had elapsed since any clinical postictal signs or symptoms (from the last observed seizure). If clinical and/or electroencephalogram monitoring showed no seizure activity, the subject received DBF single dose determined by age and body weight.
- Ictal/Peri-ictal State, Then Interictal State: The ictal/peri-ictal state was defined as an ongoing clinically observable seizure or seizure activity as verified via EEG. The peri-ictal state was defined as the subject's immediate postictal state following a generalized tonic-clonic (GTC) seizure or focal seizure with impaired awareness, and within 5 minutes after the last clonic jerk. For subjects on EEG monitoring, the peri-ictal state could be defined as less than 5 minutes after cessation of seizure activity (GTC or focal seizure with impaired awareness) as verified via EEG.
Period: Overall Study
Arm/Group | Interictal State, Then Ictal/Peri-ictal State | Ictal/Peri-ictal State, Then Interictal State
Started | 11 | 13
Completed | 3 | 6
Not Completed | 8 | 7
Not completed — Treatment B not done | 5 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Treatment A not done | 0 | 5
Not completed — Study terminated by sponsor | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: The safety analysis set comprised all subjects who received at least 1 dose of DBF determined according to the weight and age of the subject.
Groups:
- Safety Analysis Set: A total of 24 subjects were enrolled and received at least 1 dose of DBF determined based on age and weight (6 in the 2-5 years age group, 9 in the 6-11 years age group, and 9 in the 12-16 years age group).
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants] — Population: Pediatric patients with epilepsy in three age ranges (2-5 years, 6-11 years, 12-16 years) who received at least 1 dose of DBF determined by age and weight
  Participants
    <=18 years | 24
    Between 18 and 65 years | 0
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.0 (1.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 14
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 22.166 (10.1980)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time Curve (AUC) 0 to 4 Hours Post-dose
Description: AUC calculated from time 0 (dosing) to 4 hours post-dose in both Period A (interictal administration) and Period B (ictal/peri-ictal administration)
Time Frame: Time 0 (dosing), 0.25, 0.5, 1, 1.5, 2, 4 hours post-dose
Population: Subjects in the Pharmacokinetics Population who had data following dosing in both the Interictal State and the Ictal/Peri-ictal State
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Interictal State: Diazepam Buccal Film administered to epileptic patients during interictal state (Period A).
  Subjects received a single dose of DBF (range 5 to 17.5 mg) determined on the basis of the subject's age and weight using an interactive web response system during check-in for the subject's first treatment period.
- Ictal/Peri-ictal State: Diazepam Buccal Film administered to epileptic patients during ictal/peri-ictal state (Period B) Subjects received a single dose of DBF (range 5 to 17.5 mg) determined on the basis of the subject's age and weight using an interactive web response system during check-in for the subject's first treatment period.
Arm/Group | Interictal State | Ictal/Peri-ictal State
Number analyzed (Participants) | 8 | 8
hr*ng/mL | 739.33 (312.06) | 585 (377.11)

2. Primary Outcome: Area Under the Concentration Time Curve (AUC) From 0 to 2 Hours Post-dose
Description: AUC calculated from time 0 (dosing) to 2 hours post-dose in both Period A (interictal administration) and Period B (ictal/peri-ictal administration)Period A (interictal administration) and Period B (ictal/peri-ictal administration)
Time Frame: Time 0 (dosing), 0.25, 0.5, 1, 1.5, 2 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Interictal State (Period A): Diazepam Buccal Film administered to epileptic patients during interictal state (Period A) Subjects received a single dose of DBF (range 5 to 17.5 mg) determined on the basis of the subject's age and weight using an interactive web response system during check-in for the subject's first treatment period.
- Ictal/Peri-ictal State (Period B): Diazepam Buccal Film administered to epileptic patients during ictal/peri-ictal state (Period B) Subjects received a single dose of DBF (range 5 to 17.5 mg) determined on the basis of the subject's age and weight using an interactive web response system during check-in for the subject's first treatment period.
Arm/Group | Interictal State (Period A) | Ictal/Peri-ictal State (Period B)
Number analyzed (Participants) | 8 | 8
hr*ng/mL | 394.63 (192.47) | 309.34 (210.39)

3. Primary Outcome: Time When Maximum Plasma Concentration Was Observed (Tmax) 0 to 2 Hours Post-dose
Description: Tmax calculated from time 0 (dosing) to 2 hours post-dose in both Period A (interictal administration) and Period B (ictal/peri-ictal administration)
Time Frame: Time 0 (dosing), 0.25, 0.5, 1, 1.5, 2 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Interictal State (Period A) | Ictal/Peri-ictal State (Period B)
Number analyzed (Participants) | 8 | 8
hours | 1.196 (0.754) | 0.861 (0.574)

4. Primary Outcome: Time When Maximum Plasma Concentration Was Observed (Tmax) 0-4 Hours Post-Dose
Description: Tmax calculated from dosing (Time 0) to 4 hours post-dose in both Period A (interictal administration) and Period B (ictal/peri-ictal administration)
Time Frame: Time 0 (dosing), 0.25, 0.5, 1, 1.5, 2, 4 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Interictal Period (Period A); Ictal/Peri-Ictal Period (Period B): Each subject received a single dose of DBF based on the subject's age and weight.
  Diazepam Buccal Film: Subjects received a single DBF dose determined by age and body weight during the interictal state and during the ictal/peri-ictal period with at least 14 days washout between doses.
Arm/Group | Interictal Period (Period A) | Ictal/Peri-Ictal Period (Period B)
Number analyzed (Participants) | 8 | 8
hours | 1.196 (0.754) | 0.861 (0.574)

5. Primary Outcome: Observed Maximum Plasma Concentration (Cmax) 0-2 Hours
Description: Maximum observed plasma concentration measured from Time 0 to 2 hours post-dose in Period A (interictal administration) and Period B (ictal/peri-ictal administration)
Time Frame: Time 0 (dosing), 0.25, 0.5, 1, 1.5, 2 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Interictal Period (Period A) | Ictal/Peri-ictal Period (Period B)
Number analyzed (Participants) | 8 | 8
ng/mL | 296.64 (152.82) | 233.50 (141.92)

6. Primary Outcome: Observed Maximum Plasma Concentration (Cmax) From Time 0 (Dosing) to 4 Hours Post-dose
Description: Maximum observed plasma concentration from Time 0 to 4 hours post-dose in Period A (interictal administration) and Period B (ictal/peri-ictal administration)
Time Frame: Time 0 (dosing), 0.25, 0.5, 1, 1.5, 2, 4 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ictal/Peri-ictal State: Diazepam Buccal Film administered to epileptic patients during ictal-peri-ictal state (Period B) Subjects received a single dose of DBF (range 5 to 17.5 mg) determined on the basis of the subject's age and weight using an interactive web response system during check-in for the subject's first treatment period.
Arm/Group | Interictal State | Ictal/Peri-ictal State
Number analyzed (Participants) | 8 | 8
ng/mL | 296.64 (152.82) | 233.50 (141.92)

7. Secondary Outcome: Usability of Diazepam Buccal Film: Number of Subjects Who Spit Out/Moved/Chewed the Film After it Adhered (Stuck) to Buccal Mucosa During Period A and Period B.
Description: Was DBF spit out or blown out by the subject after adherence to the buccal mucosa or did the subject chew, talk or move the DBF prior to complete disintegration/dissolution?
Time Frame: Period A and Period B from the time of first attempt at DBF insertion to 15 minutes after insertion.
Population: The safety population comprising all subjects who received at least 1 dose of the study drug in the given study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Interictal Period (Period A) | Ictal/Peri-ictal Period (Period B)
Number analyzed (Participants) | 17 | 16
Participants | 3 | 1

8. Secondary Outcome: Usability of Diazepam Buccal Film: Unsuccessful Attempts
Description: Number of subjects with any unsuccessful DBF insertion attempts (All analyzed subjects with an unsuccessful attempt ultimately had a successful attempt at dosing)
Time Frame: Period A and Period B from the time of first attempt at DBF insertion to 15 minutes after insertion.
Population: The safety population comprising all subjects who received at least 1 dose of the study drug in the given study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Interictal Period (Period A) | Ictal/Peri-ictal Period (Period B)
Number analyzed (Participants) | 17 | 16
Participants | 0 | 4

9. Secondary Outcome: Usability Endpoint : Amount of Saliva That Exited the Mouth After DBF Dosing
Description: Estimation of the amount of saliva exiting the mouth in mL after DBF dosing in Period A and Period B
Time Frame: Period A and Period B from the time of first attempt at DBF insertion to 15 minutes after insertion.
Population: The safety population comprising all subjects who received at least 1 dose of the study drug in the given study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Interictal Period (Period A) | Ictal/Peri-Ictal Period (Period B)
Number analyzed (Participants) | 17 | 16
Participants
  Participants with 0 mL saliva exiting the mouth | 13 | 15
  Participants with > 0 mL to ≤ 1 mL saliva exiting the mouth | 0 | 1
  Participants with > 1 mL to ≤ 2 mL saliva exiting the mouth | 2 | 0
  Participants with > 2 mL to ≤ 3 mL saliva exiting the mouth | 1 | 0
  Participants with no data reported or unknown | 1 | 0

10. Secondary Outcome: Number of Subjects Who Swallowed DBF After Initial Insertion
Description: Number of subjects who swallowed DBF during Period A and/or Period B
Time Frame: Period A and Period B from the time of first attempt at DBF insertion to 15 minutes after insertion.
Population: The safety population comprising all subjects who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Interictal Period (Period A) | Ictal/Peri-ictal Period (Period B)
Number analyzed (Participants) | 17 | 16
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of informed consent through 14 days +/- 2 days after dosing
Arm/Group | Interictal Period (Period A) | Ictal/Peri-ictal Period (Period B)
All-Cause Mortality (participants affected / at risk) | 0/17 | 2/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 2/16
Other Adverse Events (participants affected / at risk) | 9/17 | 7/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interictal Period (Period A) (N=17) | Ictal/Peri-ictal Period (Period B) (N=16)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Seizure cluster (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interictal Period (Period A) (N=17) | Ictal/Peri-ictal Period (Period B) (N=16)
Seizure (Nervous system disorders) | 1 (1) | 3 (10) — Seizure activity was reported as adverse event
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Petit mal epilepsy (General disorders) | 1 (1) | 1 (1) — Absence seizure
Generalized tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (5) — Tonic-clonic seizure
Myoclonic epilepsy (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Headache
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) — Upper respiratory infection
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) — Pneumonia
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) — Sinus infection
Pyexia (General disorders) | 2 (2) | 1 (1) — Fever
Vomiting (Gastrointestinal disorders) | 1 (4) | 0 (0) — Vomiting
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Nausea
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Labored breathing
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Rash on upper extremity and face

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT03222349/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT03222349/SAP_001.pdf